CLINICAL TRIAL: NCT01451762
Title: A Dose Ranging Effect of Preoperative Diphenhydramine on Postoperative Quality of Recovery After Ambulatory Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Gildasio De Oliveira, Gildasio De Oliveira, M.D. Principal Investigator, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: STU00044695
Record Dates: First submitted 2011-09-20; First posted 2011-10-14 (Estimated); Results first posted 2014-03-14 (Estimated); Last update posted 2014-03-14 (Estimated); Status verified 2014-02

CONDITIONS: Surgery; Pain
Keywords: pain; anesthesia; surgery; postoperative
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Placebo (Placebo Comparator): .9 normal saline IV
  Interventions: Drug: .9 normal saline
- 25 mg diphenhydramine IV (Active Comparator): 25 mg diphenhydramine IV administered before surgery
  Interventions: Drug: 25 mg diphenhydramine IV
- 50 mg diphenhydramine IV (Active Comparator): 50 mg diphenhydramine IV administered before surgery
  Interventions: Drug: 50 mg diphenhydramine IV

INTERVENTIONS:
Drug: .9 normal saline — .9 normal saline administered before surgery.
  Arms: Placebo
Drug: 25 mg diphenhydramine IV — 25 mg diphenhydramine IV administered before surgery
  Arms: 25 mg diphenhydramine IV
Drug: 50 mg diphenhydramine IV — 50 mg diphenhydramine administered IV before surgery
  Arms: 50 mg diphenhydramine IV

SUMMARY:
Pain after ambulatory surgery remains an unsolved problem in The United States and Europe. It is associated with delayed hospital discharge and it can result to an increased opioid consumption with adverse side effects. The concept of multimodal analgesic technique was introduced more than 15 years ago and several techniques have been studied over the years including non steroidal antiinflammatory drugs (NSAIDs), acetaminophen, gabapentoids, ketamine, local and regional anesthetic techniques. Histamine can have effects on polymodal nociceptors and C-fibers, producing pain which is further increased by neurogenically mediated release of substance P from afferent pain fibers. Several non-selective or H1 -selective histamine receptors antagonists have been demonstrated in animal models and clinical pain. Chia et al demonstrated that preoperative promethazine had opioid sparing properties without adverse sedative effects in patients undergoing abdominal hysterectomy.

Diphenhydramine is an anti-histamine drug who has been found to be effective in reducing postoperative nausea and vomiting after ambulatory surgery but its effects on postoperative pain and other important outcomes after ambulatory surgery such as time to meet discharge criteria have not being studied.

The MQOR 40 is a validated instrument that was specifically design to evaluate patient recovery after anesthesia and surgery. This instrument can be particularly valid to examine interventions which affect different spheres of patient recovery as is the case of diphenhydramine. The objective of this study is to determine a dose response effect of preoperative diphenhydramine on postoperative quality of recovery after ambulatory surgery. The use of preoperative diphenhydramine can improve patient's quality of recovery, decrease postoperative pain, opioid consumption and opioid related side effects after ambulatory surgery.

The research question: Does a preoperative dose of diphenhydramine improve postoperative quality of recovery after ambulatory surgery? The hypothesis of this study is that preoperative diphenhydramine will improve postoperative pain, Postoperative nausea and vomiting (PONV), sleep which will translate in a better overall quality of recovery.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-64 years
* Patients undergoing ambulatory surgery
* ASA PS I, II.

Exclusion Criteria:

* Chronic opioid use
* pregnant patient or lactating patients
* allergy to diphenhydramine
* glaucoma
* uncontrolled hypertension
* asthma
* hyperthyroidism
* cardiovascular disease

Ages: 18 Years to 64 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2011-09; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gildasio De Oliveira, MD, Principal Investigator — Northwestern University
Locations (2):
- United States (2):
  - Prentice Womens HOspital, Chicago, Illinois
  - Prentice Womens HOsptial, Chicago, Illinois

REFERENCES:
- [Background] Apfelbaum JL, Chen C, Mehta SS, Gan TJ. Postoperative pain experience: results from a national survey suggest postoperative pain continues to be undermanaged. Anesth Analg. 2003 Aug;97(2):534-540. doi: 10.1213/01.ANE.0000068822.10113.9E. PMID 12873949
- [Background] Benhamou D, Berti M, Brodner G, De Andres J, Draisci G, Moreno-Azcoita M, Neugebauer EA, Schwenk W, Torres LM, Viel E. Postoperative Analgesic THerapy Observational Survey (PATHOS): a practice pattern study in 7 central/southern European countries. Pain. 2008 May;136(1-2):134-41. doi: 10.1016/j.pain.2007.06.028. Epub 2007 Aug 20. PMID 17703887
- [Background] Kehlet H, Dahl JB. The value of "multimodal" or "balanced analgesia" in postoperative pain treatment. Anesth Analg. 1993 Nov;77(5):1048-56. doi: 10.1213/00000539-199311000-00030. No abstract available. PMID 8105724
- [Background] White PF, Kehlet H. Improving postoperative pain management: what are the unresolved issues? Anesthesiology. 2010 Jan;112(1):220-5. doi: 10.1097/ALN.0b013e3181c6316e. No abstract available. PMID 20010418
- [Background] Schmelz M, Schmidt R, Bickel A, Handwerker HO, Torebjork HE. Specific C-receptors for itch in human skin. J Neurosci. 1997 Oct 15;17(20):8003-8. doi: 10.1523/JNEUROSCI.17-20-08003.1997. PMID 9315918
- [Background] Baird-Lambert J, Jamieson DD. Possible mediators of the writhing response induced by acetic acid or phenylbenzoquinone in mice. Clin Exp Pharmacol Physiol. 1983 Jan-Feb;10(1):15-20. doi: 10.1111/j.1440-1681.1983.tb00166.x. PMID 6188566
- [Background] Rumore MM, Schlichting DA. Analgesic effects of antihistaminics. Life Sci. 1985 Feb 4;36(5):403-16. doi: 10.1016/0024-3205(85)90252-8. PMID 2578597
- [Background] Raffa RB. Antihistamines as analgesics. J Clin Pharm Ther. 2001 Apr;26(2):81-5. doi: 10.1046/j.1365-2710.2001.00330.x. PMID 11350529

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 90 subjects were enrolled between September 2011 and September 2012.
Period: Overall Study
Arm/Group | Placebo | 25 mg Diphenhydramine IV | 50 mg Diphenhydramine IV
Started | 30 | 30 | 30
Completed | 27 | 24 | 24
Not Completed | 3 | 6 | 6
Not completed — Lost to Follow-up | 3 | 6 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | 25 mg Diphenhydramine IV | 50 mg Diphenhydramine IV | Total
Number analyzed (Participants) | 30 | 30 | 30 | 90
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 30 | 30 | 30 | 90
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 35 (8.36) | 36.5 (10.7) | 37 (8.3) | 37 (9.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 30 | 30 | 90
  Male | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 30 | 30 | 30 | 90

OUTCOME MEASURES:

1. Primary Outcome: Quality of Recovery 40 at 24 Hours
Description: Scores on QOR (quality of recovery) 40 questionnaire.The QoR-40 score, which ranges from 40 to 200, representing very poor to outstanding quality of recovery, respectively.
Time Frame: 24 hours post operatively
Population: Primary outcome was QOR 40 a sample size of 23 per group was estimated to achieve 80% power to detect a 10 point difference in aggregated QOR040 score for the three groups. A 10 point difference represents a clinically relevant improvement in quality of recovery. TO account for drop outs lost to follow up 90 subjects were randomized.
Measure: Median (Inter-Quartile Range); unit: units on scale 40 (low) - 200 (high)
Arm/Group | Placebo | 25 mg Diphenhydramine IV | 50 mg Diphenhydramine IV
Number analyzed (Participants) | 27 | 24 | 24
units on scale 40 (low) - 200 (high) | 164 [151 to 189] | 169 [159 to 181] | 172 [157 to 185]

ADVERSE EVENTS:
Time Frame: 24 hours
Arm/Group | Placebo | 25 mg Diphenhydramine IV | 50 mg Diphenhydramine IV
Serious Adverse Events (participants affected / at risk) | 0/27 | 0/24 | 0/24
Other Adverse Events (participants affected / at risk) | 12/27 | 9/24 | 3/24
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=27) | 25 mg Diphenhydramine IV (N=24) | 50 mg Diphenhydramine IV (N=24)
Nausea (Gastrointestinal disorders) | 12 (12) | 9 (9) | 3 (3)

LIMITATIONS AND CAVEATS:
We did not obtain preoperative quality of recovery scores of patients therefore we could not examine whether the effect of diphenhydramine was dependent upon patient's baseline characteristics.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No